CLINICAL TRIAL: NCT00998153
Title: Risk Reduction for Drug Use and Sexual Revictimization
Acronym: RRFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DA018686 (NIH); K23DA018686 (NIH)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Risk Reduction Through Family Therapy; Usual Care
Keywords: substance use; PTSD; risky behaviors; revictimization
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): RRFT
  Interventions: Behavioral: Risk Reduction through Family Therapy
- 2 (Active Comparator): Usual care
  Interventions: Behavioral: Risk Reduction through Family Therapy

INTERVENTIONS:
Behavioral: Risk Reduction through Family Therapy — Component based intervention based on existing empirically supported treatments
  Other Names: RRFT

SUMMARY:
The investigator proposes to evaluate Risk Reduction through Family Therapy (RRFT), which integrates: 1) an ecologically-based intervention for treatment of substance abuse behaviors in high risk adolescents, 2) exposure-based cognitive-behavioral therapy for sexually assaulted youth, and 3) psychoeducation strategies for prevention of risky sexual behaviors and revictimization. The principal purpose of this research proposal is to evaluate the efficacy of RRFT in reducing the risk of drug abuse and other risky behaviors, PTSD, and revictimization among adolescents who have been sexually assaulted. The Research Plan will be conducted based on Stage 1a and Stage 1b from NIDA's Behavioral Therapies Development Program as described in Rounsaville, Carroll, & Onken (2001). The final phase of the research will involve conducting a pilot randomized controlled trial of RRFT in a sample of adolescents, comparing primary outcome measures of youth receiving RRFT to youth receiving usual care in the community. Participants will be adolescents (12-17 years) who have experienced a sexual assault. Assessment of substance use and other risk behaviors, trauma-related psychopathology, and incidents of revictimization will be collected at pre- and post- treatment, as well as 6-week and 3-month follow-ups. Hierarchical Linear Modeling will be the primary method used to test study hypotheses. Development and evaluation of the proposed intervention will have significant implications for addressing public health problems in adolescent substance abuse and related high risk behaviors.

DETAILED DESCRIPTION:
See above summary

ELIGIBILITY:
Inclusion Criteria:

* memorable sexual assault

Exclusion Criteria:

* active psychosis
* active suicidality

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2012-06-30 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back and urine screen | Pre and post-treatment, 3 and 6 month follow-ups

SECONDARY OUTCOMES:
YRBS | Pre and post-treatment, 3 and 6 month follow-ups
FES | Pre and post-treatment, 3 and 6 month follow-ups
UCLA PTSD Reaction Index | Pre, post, and 3 and 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Crime Victims Research and Treatment Center, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Danielson CK, McCart MR, Walsh K, de Arellano MA, White D, Resnick HS. Reducing substance use risk and mental health problems among sexually assaulted adolescents: a pilot randomized controlled trial. J Fam Psychol. 2012 Aug;26(4):628-35. doi: 10.1037/a0028862. Epub 2012 Jun 11. PMID 22686269